CLINICAL TRIAL: NCT07182396
Title: Effects of Video Games and Ball Tossing on Eye Hand Coordination in Elderly With Mild Cognitive Impairment.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/04
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Dysfunction; Cognitive Disorder; Cognitive Decline
Keywords: Eye hand coordination; mild cognitive impairment; video games intervention; MoCA; Beery VMI( Beery Buktenica developmental test)
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video games and ball tossing intervention (Experimental): TAPD game:Tap the correct targets as they scroll down the screen. Be careful, though, the current target colour will change and the scrolling speed will increase progressively by time. it will have 5 difficulty levels Hand eye coordination game:Tap changing illuminating squares
  Ball tossing intervention:
  Exercise 1: Participant will be supposed to dribble/ tap soft bouncing ball on ground with one hand. After one set of exercise, 2 minutes of rest will be given and then again same exercise will be performed.
  Exercise 2: Participants will be supposed to throw soft ball to the wall and aim for re-bound catch, initially starts from football sized soft ball and progress to small ball to increase difficulty level according to participants.
  For easy level, participants can start from catching the ball after tapping to ground in the first week depending upon their ability.
  Exercise 3: Participants will be supposed to tap table tennis ball with table tennis bat in air in vertical direction
  Interventions: Procedure: Experimental Group
- ball tossing intervention (Active Comparator): Exercise 1: Participant will be supposed to dribble/ tap soft bouncing ball on ground with one hand. After one set of exercise, 2 minutes of rest will be given and then again same exercise will be performed.
  Exercise 2: Participants will be supposed to throw soft ball to the wall and aim for re-bound catch, initially starts from football sized soft ball and progress to small ball to increase difficulty level according to participants.
  For easy level, participants can start from catching the ball after tapping to ground in the first week depending upon their ability.
  Exercise 3: Participants will be supposed to tap table tennis ball with table tennis bat in air in vertical direction
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Experimental Group — VIDEO GAME-TAPD: Week 1st-6th: Start with kids level and progress upto expert level and Participants will automatically progress to advanced level based on their individual ability and progress in game in progressing weeks.
  (kids level to expert level: according to game levels) Hand eye coordination game:Tap changing illuminating squares. Week1- 3 repetitions(2sets),Week2- 4 repetitions(2 sets),Week3- 5 repetitions(2 sets),Week4- 6 repetitions(2 sets),Week5- 7 repetitions(2 sets),Week6- 8 repetitions(2 sets) Ball tossing intervention:Week 1-2 (Exercise 1 (2 sets, 20/30/40 repetitions) and Exercise 2(2 sets, 20/30/40 repetitions) with ground tap catch Week 3-4 (Exercise 2 (2 sets, 20/30/40 repetitions) with direct catch and Exercise 3 (2 sets, 20/30/40 repetitions) Week 5-6 (Exercise 1 (2 sets, 50 repetitions) , Exercise 2 (2 sets, 50 repetitions) with direct catch and Exercise 3 (2 sets, 50 repetitions) Number of reps adjusted according to session number per week
  Arms: video games and ball tossing intervention
Procedure: Control Group — Week 1-2 (Exercise 1 (2 sets, 20/30/40 repetitions) and Exercise 2(2 sets, 20/30/40 repetitions) with ground tap catch Week 3-4 (Exercise 2 (2 sets, 20/30/40 repetitions) with direct catch and Exercise 3 (2 sets, 20/30/40 repetitions) Week 5-6 (Exercise 1 (2 sets, 50 repetitions) , Exercise 2 (2 sets, 50 repetitions) with direct catch and Exercise 3 (2 sets, 50 repetitions) Number of reps adjusted according to session number per week e.g
  * Day 1: 20 reps per week
  * Day 2: 30 reps per week
  * Day 3: 40 reps per week Progression: Participants will progress to advanced level based on their individual ability and progress. Levels of complexity will be adjusted according to patient progress.
  Arms: ball tossing intervention

SUMMARY:
One of the key challenges faced by individuals with mild cognitive impairment (MCI) is the decline in cognitive and motor abilities, particularly eye-hand coordination (EHC), which is essential for performing daily activities and maintaining independence. Impaired EHC can severely affect the quality of life in older adults, leading to difficulties in performing routine tasks like dressing, eating, and bathing, and increasing dependency on caregivers.

Signs and symptoms include difficulty with precise movements like buttoning clothes, spilling drinks while pouring, struggling to catch a ball, messy handwriting. This study aims to explore and compare the effectiveness of two interventions-video games and ball tossing exercises-in improving Eye-hand coordination (EHC) in older adults with Mild Cognitive Impairment (MCI).

Key outcome measures, including the Beery-Buktenica Developmental Test of Visual-Motor Integration (Beery VMI) and its supplemental test visual perception test and motor coordination test, will evaluate the effectiveness of the interventions on eye hand coordination.

We will include older adults with 60 and above age with MoCA score of 18-25(MCI patients), who can do independent ADLs and beery vmi score of 80 and above.

The participants would be assessed at the start of intervention through MoCA scale for MCI screening and Beery VMI testing method for Eye Hand Coordination for inclusion score.

DETAILED DESCRIPTION:
A reduction in cognitive function that occurs during the transitional period from normal aging to dementia is known as mild cognitive impairment (MCI) As people age, they experience a decline in cognitive function.The overall prevalence of MCI was 15.56% in older aged people.

Older individuals with MCI, they commonly face a decline in both cognitive and motor abilities, which can severely affect their quality of life.

One of the consequence of cognitive decline is impaired hand-eye coordination, a critical skill for daily activities and maintaining independence This impairment arises as MCI affects cognitive functions such as attention, making it difficult for individuals to focus on tasks, often leading to wandering hand and eye movements and hesitation during actions.

Hand-eye coordination, the brain's ability to synchronize visual input with hand movements, plays an essential role in performing activities of daily living (ADLs) and independence of older adults. Impaired hand-eye coordination is associated with the early stages of cognitive decline, indicating that cognitive deterioration has a significant impact on this ability.

Signs and symptoms include difficulty with precise movements like buttoning clothes, spilling drinks while pouring, struggling to catch a ball, messy handwriting, clumsiness when reaching for objects, frequent misjudging distances, and taking longer to complete tasks requiring hand-eye coordination due to slower reaction times etc.

Older adults with MCI are at risk of further cognitive decline which can lead to dementia/Alzheimer's disease in which hand-eye coordination may decline so easy, accessible and engaging intervention for older adults that will improve hand eye coordination will be provided in this study.

This study aims to determine the effect of two such interventions-video games and ball tossing exercises-in enhancing eye-hand coordination in older adults with mild cognitive impairment. This study aims to determine the effect of two such interventions-video games and ball tossing exercises-in enhancing eye-hand coordination in older adults with mild cognitive impairment.

By exploring the effects of these two interventions, this research seeks to contribute valuable insights for health care professionals to engage older population into targeted activities so they can support the cognitive health of older adults, ultimately improving their quality of life and limiting the effects of MCI like impaired eye hand coordination.

one control group will undergo exercise program only and another experimental group will play video games to improve eye hand coordination along with exercise plan A randomized control trial was conducted in 2023 on efficacy of multi-domain cognitive function training on cognitive function, working memory, attention, and coordination in older adults with mild cognitive impairment and mild dementia in which the MCFT intervention showed positive effects in enhancing global cognitive function, and hand eye coordination in older adults with mild cognitive impairment Another study in 2020 was conducted in which Analysis of a Video Game on Cognitive Abilities: A Study to Enhance Psychomotor Skills via Game-Play in which the study's findings indicate that participants aged (16-19) who played the video game showed greater confidence in their eye-hand coordination and visual responses.

They were able to complete the natural building block task more quickly and accurately A randomized control trial was conducted in 2019 in which Effect of interactive cognitive-motor training on eye-hand coordination and cognitive function in older adults was seen results show The visual-motor integration results showed a small to moderate effect size for pre post comparison A study was conducted in 2018 in students of mean age (17-18 years) and the results showed significant improvement of Hand-eye coordination compare to control group after the 4 weeks of exercise program. Experimental group performed specific exercises(bouncing ball taps and tennis ball tapping)weekly twice for four weeks In study of 2019, Results of a study suggest that playing an easily accessible video game in older age can enhance cognitive functioning, especially in areas directly tied to the video gaming activities.

This highlights the importance of identifying interventions that may help improve hand-eye coordination in older adults with MCI, thereby promoting independence and improving their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Older population aged from 60years and above
* Normal/ normal to corrected vision
* MoCA Score of 18-25 for screening / MCI patients
* Can do Independent ADLS
* Beery VMI Score: 80 and above score

Exclusion Criteria:

* History of head trauma, loss of consciousness, stroke, rapid cognitive decline
* Diagnosis of mental illness/neurocognitive disorders
* Diagnosed Vestibular disorders
* Hearing, vision and communication impairments

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
VISUAL-MOTOR INTEGRATION | 6 weeks
  The Beery-Buktenica Developmental Test of Visual-Motor Integration (Beery VMI) is a gold standard measure designed to identify challenges related to the coordination of visual and motor skills like eye hand coordination in both children and adults aged (2-100) year old.
  Visual Motor Integration takes approximately 10-15 min. Raw scores on the Beery VMI can range from 1 to 27, with a higher score reflecting a better performance.
  Raw scores are converted into standard scores according to age and each part of test has total of 30 scores to mark as there are 30 each shapes/tasks to complete.
  Interpretation:
  Standard Score Range & Interpretation:
  >129 = Very high 120-129 = High 110-119 = Above average 90-109 = Average 80-89 = Below average 70-79 = Low

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan